CLINICAL TRIAL: NCT04372316
Title: The Efficacy of Mecobalamin Injection and Tablet Treatment on Mild to Moderate Diabetic Peripheral Neuropathy： a Randomized Controlled Clinical Trial
Brief Title: A Randomized Controlled Trial of Mecobalamin Injection and Tablet Treatment Efficacy on Mild to Moderate Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Fan Dongsheng, Director, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUTH2017286
Record Dates: First submitted 2020-04-26; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — mecobalamin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylcobalamin injection (Active Comparator)
  Interventions: Drug: methylcobalamin
- methylcobalamin tablet (Active Comparator)
  Interventions: Drug: methylcobalamin

INTERVENTIONS:
Drug: methylcobalamin — methylcobamin injection 8 weeks or tablet 8 weeks， followed by 24 weeks methylcobamin tablet until 32 weeks

SUMMARY:
To evaluate the efficacy of mecobalamin injection and tablet in the treatment of small fiber lesions in the early stage of diabetic peripheral neuropathy by corneal confocal microscopy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 1 or 2 diabetes for at least 1 year
* must be consistent with the diagnosis of distal, symmetrical, sensorimotor polyneuropathy
* according to the clinical judgment of the researchers, the blood glucose has been under the best control. Before screening visit, HbA1c level ≤ 9%. During the course of the study, the blood glucose was adjusted under the guidance of the researchers, and the blood glucose was kept stable as much as possible.
* Toronto clinical neuropathy score (TCSs) ≤ 5 at screening visit
* no history of eye injury and laser treatment
* no history of keratopathy or other intraocular and extraocular diseases
* no wearing history of corneal contact lens
* no drugs affecting corneal metabolism
* no Mecobalamin or lipoic acid in 3 months
* women of childbearing age (e.g. non-surgical contraception or menopause less than 1 year) must be negative in the gonadotropin pregnancy test (urine) during the screening period, and effective contraceptive measures must be taken during the treatment period and within 1 month after the end of the treatment
* the participant signs the informed consent, indicating that the subject has been informed of all research related contents
* participants are willing and able to follow study visit arrangements, treatment plans, laboratory tests and other research procedures

Exclusion Criteria:

* has been diagnosed as a malignant tumor in the past 2 years.
* the presence of other neurological disorders that the researchers believe may affect the evaluation of diabetic peripheral neuropathy
* presence of skin disease in the affected skin area, which, in the judgment of the researchers, may affect the evaluation of diabetic peripheral neuropathy
* amputations other than finger ends and toes
* participated in any other studies or post market drugs studies within 30 days prior to screening
* participants with clinically significant or unstable diseases, such as but not limited to acute cardiovascular disease, cerebrovascular disease, liver, kidney, respiratory system, blood system, immune system, inflammatory or rheumatic disease, uncontrolled infection, symptomatic peripheral vascular disease, untreated endocrine disease, etc
* have donated blood within 30 days prior to the start of the study treatment (if applicable); or have prepared blood donors during the study or within 30 days after the end of the treatment
* WBC < 4000 / mm3; neutrophil count < 1500 / mm3; platelet count < 100 × 103 / mm3
* clinically significant abnormal 12 lead ECG
* participants received combined transcutaneous electrical nerve stimulation (TENS) or acupuncture
* previous history of intolerance or allergies to study drugs or drugs with similar chemical structure
* has a history of alcohol and / or other drug abuse in the past year or is currently under the influence of alcohol or drug abuse
* the presence of other acute or chronic medical or psychiatric conditions or laboratory abnormalities that, in the judgment of the investigator, may increase the risk associated with participating in the trial or using the study product, or may affect the interpretation of the study results, may make the subject unsuitable for the trial
* inability and / or unwillingness to understand and / or comply with the program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-25 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
changes of inferior whorl length （IWL）from baseline at 8 weeks | 8 weeks
  changes of the nerve length of inferior whorl area of each mm2

SECONDARY OUTCOMES:
changes of corneal nerve fiber length（CNFL）from baseline at 8 weeks | 8 weeks
  changes of corneal nerve fiber length sum of each mm2
changes of corneal nerve branch density（CNBD）from baseline at 8 weeks | 8 weeks
  changes of corneal nerve branch density of each mm2
changes of corneal nerve fibre density（CNFD）from baseline at 8 weeks | 8 weeks
  changes of corneal nerve fibre density of each mm2
changes of corneal nerve fibre tortuosity （CNFT) from baseline at 8 weeks | 8 weeks
  changes of corneal nerve fibre tortuosity

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang Y, Fan D, Zhang Y, Zhang S, Wang H, Liu Z, Wang H. Using corneal confocal microscopy to compare Mecobalamin intramuscular injections vs oral tablets in treating diabetic peripheral neuropathy: a RCT. Sci Rep. 2021 Jul 19;11(1):14697. doi: 10.1038/s41598-021-94284-4. PMID 34282267